CLINICAL TRIAL: NCT03738332
Title: Low-Level Laser in Treatment of Head and Neck Lymphedema: A Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Jie Deng, Associate Professor, PhD, University of Pennsylvania
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: UPCC12318
Record Dates: First submitted 2018-11-08; First posted 2018-11-13 (Actual); Results first posted 2022-01-25 (Actual); Last update posted 2022-02-01 (Actual); Status verified 2022-01

CONDITIONS: Head and Neck Cancer; Lymphedema; Fibrosis
MeSH Terms: conditions — Head and Neck Neoplasms; Lymphedema; Fibrosis | interventions — Low-Level Light Therapy

STUDY DESIGN:
Intervention Model Description: Pre-and post design
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Low-level laser therapy (Other): Single arm
  Interventions: Device: Low-Level Laser

INTERVENTIONS:
Device: Low-Level Laser — Low-level laser therapy

SUMMARY:
The purpose of this pilot clinical trial is to evaluate the feasibility of the use of low-level laser for head and neck cancer survivors with lymphedema.

DETAILED DESCRIPTION:
Primary aim:

To determine the feasibility of the use of LLLT for HNC survivors with lymphedema, specifically to 1) obtain recruitment estimates and determine barriers to recruitment; 2) identify barriers to implementation; 3) assess safety; and 4) evaluate patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* >18 years of age
* Completion of either postoperative radiation or chemoradiation therapy
* No evidence of cancer
* Having head and neck external lymphedema
* Either completion of lymphedema therapy or not in active lymphedema therapy
* Ability to speak and read English
* Able to provide informed consent

Exclusion Criteria:

Patients will be excluded if they have any of the following medical conditions that would prohibit the safe implementation of LLLT: pregnancy; photosensitivity; chronic inflammatory diseases; venous thrombosis; history of severe trauma; medication that affects body fluid and electrolyte balance; use of high doses of non-steroidal anti-inflammatory drugs; or pre-existing skin rash, ulceration, open wound in the treatment area; and allergic and other systemic skin diseases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-02-25 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania Abramson Cancer Center, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Deng J, Lukens JN, Zhu J, Cohn JC, Andersen LP, Spinelli BA, Quinn RJ, Chittams J, McMenamin E, Lin A. Patient Experience of Photobiomodulation Therapy in Head and Neck Chronic Lymphedema. J Palliat Med. 2023 Sep;26(9):1225-1233. doi: 10.1089/jpm.2021.0419. Epub 2023 Apr 28. PMID 37116057
- [Derived] Deng J, Lukens JN, Swisher-McClure S, Cohn JC, Spinelli BA, Quinn RJ, Chittams J, McMenamin E, Lin A. Photobiomodulation Therapy in Head and Neck Cancer-Related Lymphedema: A Pilot Feasibility Study. Integr Cancer Ther. 2021 Jan-Dec;20:15347354211037938. doi: 10.1177/15347354211037938. PMID 34387119

RESULTS

PARTICIPANT FLOW:
Groups:
- Low-level Laser Therapy: Single arm
  Low-Level Laser: Low-level laser therapy Dose: twice a week for 6 weeks (12 sessions)
Period: Overall Study
Arm/Group | Low-level Laser Therapy
Started | 12
Completed | 11
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Low-level Laser Therapy
Number analyzed (Participants) | 12
Age, Continuous [Mean (Full Range); unit: years] | 58.4 [32 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 11
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Consented and Enrolled in Study
Description: Number of participants who consented the study and number of participants who enrolled in the study
Time Frame: Approximately 5-month recruitment window
Measure: Count of Participants; unit: Participants
Arm/Group | Low-level Laser Therapy
Number analyzed (Participants) | 30
Participants | 12

2. Primary Outcome: Number of Participants Completed the Study Visits
Description: Number of participants who completed the study visits
Time Frame: Approximately 10 weeks, from baseline visit to 4-week post-intervention visit
Measure: Count of Participants; unit: Participants
Arm/Group | Low-level Laser Therapy
Number analyzed (Participants) | 12
Participants | 11

3. Primary Outcome: Number of Participants With Adverse Events
Description: Number of participants who experienced adverse events during the course of the study.
Time Frame: Approximately 10 weeks, from baseline visit to 4-week post-intervention visit
Measure: Count of Participants; unit: Participants
Arm/Group | Low-level Laser Therapy
Number analyzed (Participants) | 12
Participants | 0

4. Primary Outcome: Number of Participants Who Were Satisfied With Study Intervention.
Description: Participants were interviewed by the study staff to ask whether they were satisfied or unsatisfied with the study intervention (low-level laser therapy).
Time Frame: at 4-week post-intervention visit
Measure: Count of Participants; unit: Participants
Arm/Group | Low-level Laser Therapy
Number analyzed (Participants) | 11
Participants | 11

ADVERSE EVENTS:
Time Frame: The adverse events were monitored and assessed during the course of the study, that is, from the start of the intervention up to 4 weeks post intervention, up to approximately 10 weeks. .
Arm/Group | Low-level Laser Therapy
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-15): https://cdn.clinicaltrials.gov/large-docs/32/NCT03738332/Prot_SAP_001.pdf